CLINICAL TRIAL: NCT00508456
Title: A Phase I Study of Dietary Methionine Restriction and Temodar® (Temozolomide) for the Treatment of Recurrent and Progressive Glioblastoma Multiforme
Brief Title: Dietary Methionine Restriction Plus Temozolomide for Recurrent GBM
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID03-0066
Record Dates: First submitted 2007-07-27; First posted 2007-07-30 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma Multiforme; Methionine Restriction; Hominex-2; Methionine Restriction Diet; Hominex-2 Amino Acid-Modified Medical Food; Temozolomide; Temodar
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hominex®-2 + Temodar® (Experimental): Dietary Methionine Restriction (Hominex®-2) Days 1-7 and 15-21 + Temodar® 150 mg/m^2 orally Days 8-15
  Interventions: Drug: Temodar (Temozolomide); Dietary Supplement: Hominex-2

INTERVENTIONS:
Drug: Temodar (Temozolomide) — 150 mg/m^2 orally once a day for 7 consecutive days (days 8 through 15).
Dietary Supplement: Hominex-2 — Methionine free diet during Days 1 - 7 and Days 15 - 21 by consuming only "shakes" containing Hominex-2®.
  Other Names: Hominex-2® shakes; Methionine restriction diet; Hominex®-2 Amino Acid-Modified Medical Food

SUMMARY:
Objectives:

1. To determine the safety, tolerability and efficacy of dietary methionine restriction for 7 days alternating with Temodar® (Temozolomide) given once a day for seven days and this repeated for up to one year in the treatment of patients with recurrent and/or progressive glioblastoma.
2. To determine the short- and long-term toxicity of dietary methionine restriction combined with Temodar® in glioblastoma patients.
3. To measure and correlate patients' tumor responses and progression-free survival with: serum methionine and peripheral blood lymphocyte methylation levels. In any patient undergoing surgery, to measure tumor alkylguanyl transferase (AGT) and methionine levels and compare to control specimens.

DETAILED DESCRIPTION:
Methionine is an essential amino acid. Many solid tumors depend on the methionine that is taken in through the diet. The tumors need methionine to grow. A methionine free (or reduced) diet may help to shrink or slow the growth of some tumors. Temozolomide is a drug that is commonly used in the treatment of glioma. A methionine free (or reduced) diet may increase the effectiveness of temozolomide in the treatment of glioma.

Before treatment, you will have a complete physical exam and blood (around 2 tablespoons) will be collected for routine tests. You will have either a magnetic resonance imaging (MRI) scan or a computed tomography (CT) scan of the brain. Women who are able to have children must have a negative blood pregnancy test. You will then meet with a study dietician. The dietician will give you written instructions and make a food plan based on your needs. The instructions and food plan will help you maintain a methionine-free (or reduced) diet during the study.

During the study, all participants will receive standard chemotherapy with temozolomide by mouth once a day at bedtime for 7 days on Days 8 through 14 and 22 through 28, every 28 days, 4 weeks This 4-week period is called a cycle of chemotherapy. This 4 week cycle will be repeated as long as the disease does not get worse.

During treatment, you will be asked to maintain a methionine free diet during Days 1 - 7 and Days 15 - 21. During the periods of methionine free diet, you will consume only "shakes" containing Hominex-2®. The Hominex-2® shakes are nutritionally complete and easy to prepare. You will be given instructions on how to maintain this methionine-free diet.

All participants enrolled in the study will consume a methionine free diet for 1 week, alternating with temozolomide chemotherapy for 1 week. The participants will then be switched to a methionine "replete" diet for 1 week while taking chemotherapy. This diet and chemotherapy schedule will be continued for as long as the treatment is effective and tolerable. This replete diet contains methionine. The dietician will record what you eat to make sure you are eating the right amount of methionine during this period. This 4-week schedule will be repeated as long as you are on the study.

If you experience any intolerable side effects or the disease gets worse, you will be taken off the study and your doctor will discuss other treatment options with you.

During treatment, you will have blood (around 1 tablespoon) collected every 2 weeks for routine tests. Every 4 weeks for the first 16 weeks then every 8 weeks for the rest of the study, you will have check up visits. At these visits, you will have a complete physical exam and have blood collected (around 1 tablespoon) for routine tests. You will also have a dietary consultation. Every 8 weeks during the study, you will have either a MRI scan or a CT scan of the brain. If your doctor feels it is necessary, the tests may be done more often or you may have other tests as needed for your care.

This is an investigational study. Methionine restriction diet (Hominex®-2 Amino Acid-Modified Medical Food) has been approved by the FDA for nutrition support of children and adults with vitamin B6-nonresponsive homocystinuria. However, its use in this study is investigational. Temozolomide has been approved by the FDA for the treatment of brain tumors and is commercially available. The use of this combination is experimental. Forty-four participants will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven glioblastoma multiforme (GBM).
2. Unequivocal evidence of tumor recurrence or progression by MRI (or CT brain if a patient can not undergo MRI). Radiotherapy (with or without radiosensitizing drugs) must have been completed in the past. The earliest a patient can be enrolled in this study after radiotherapy is 14 days. The scan done prior to study entry documenting progression will be reviewed by the primary investigator to document tumor volume changes to provide a gross assessment of growth rate.
3. Patients may have had: a) no prior chemotherapy, b) 1 prior adjuvant chemotherapy, c) 1 prior adjuvant chemotherapy followed by 1 regimen for recurrent disease, or d) 1 or 2 prior chemotherapy regimens for recurrent or progressive tumor.
4. All patients must sign an informed consent indicating that they are aware of the investigational nature of this study in keeping with the policies of this hospital.
5. Enrollment MRI or CT scan of the brain must be performed within 14 days of registration. Patients having undergone recent resection of recurrent or progressive tumor will be eligible for assessment of response as long as there is residual enhancing evaluable disease that is documented by appropriate neuroimaging and patients have recovered from the effects of surgery. Patients who after surgery have no residual enhancing disease will still be eligible for enrollment, but only assessable for time to progression, and not for response.
6. Patients must have a life expectancy > 8 weeks.
7. Patients must have a Karnofsky performance status of > or = 60 (Karnofsky Performance Scale).
8. Patients must have recovered from the toxic effects of prior therapy and/or at least 2 weeks from vincristine, 6 weeks from nitrosoureas, and 3 weeks from procarbazine administration. Patients must have recovered from the toxic effects of any other cytotoxic drugs which they may have received and must be 1 week from the completion of any non-cytotoxic drug therapy (e.g. 13-cis-retinoic acid, thalidomide, tamoxifen, etc.). For those patients previously treated with temozolomide, they may enroll and start the diet even 1 day after their last temozolomide dose.
9. Patients must have adequate bone marrow function (ANC> or = 1,500/mm3 and platelet count of > or = 100,000/mm3), adequate liver function (SGPT and alkaline phosphatase = or <2 times normal, bilirubin = or <1.5 mg%), and adequate renal function (BUN or creatinine = or <1.5 times institutional normal) prior to starting therapy.
10. All acute toxic effects (excluding neurotoxicity or alopecia) of any prior therapy must have resolved to Common Toxicity Criteria (CTC) grade = or < 1.
11. Patients who are eligible for the trial and who require resection of their tumor may begin the dietary restriction component of the therapy prior to their surgery providing the time to surgery is greater than 6 days. In these patients, tissue collected at surgery will be analysed for the effects of treatment. After surgery, patients will resume an ad lib diet for anywhere from 5-14 days prior to the re-initiation of the dietary methionine restriction at the same dose level and continuance with the trial.

Exclusion Criteria:

1. Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years.
2. Patients have one or more of the following conditions may not participate in this study: a) active infection; b) pregnancy and/or disagree to practice adequate contraception; c) disease that will obscure toxicity or dangerously alter drug metabolism; d) serious intercurrent medical illness.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Time to Disease Progression | 6 months (26 weeks)
  Time to progression measured from the first day of treatment until progression is documented.

CONTACTS AND LOCATIONS:
Overall Officials: Morris D. Groves, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org